CLINICAL TRIAL: NCT00446576
Title: A Study in Early Renal Insufficiency Patients to Assess the Effect of Maintaining Three Different Hemoglobin Levels With the Use of Erythropoetin Alpha on Left Ventricular Hypertrophy and Dilation and Quality if Life; The "Cardiac Results of Early Treatment of Anaemia (CRETA)" Study
Brief Title: The Effect of Epoetin Alfa on Cardiac Function and Quality of Life in Patients With Early Renal ((Kidney) Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag B.V. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005599
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Anemia
Keywords: Anemia; early renal insufficiency
MeSH Terms: conditions — Anemia; Renal Insufficiency | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
The purpose of this study is to assess whether maintaining hemoglobin (Hb) levels at normal or sub-normal levels with Epoetin Alfa can influence the health status, left ventricular mass and quality of life of early renal insufficiency subjects without additional safety concerns.

DETAILED DESCRIPTION:
The use of Epoetin alfa in the treatment of anaemia in chronic renal failure (CRF) patients is well accepted. The severity of anaemia in CRF patients increases with the degree of renal dysfunction. Thus, the most severe degree of anaemia is generally found in patients with end stage renal disease who must be maintained on dialysis. Nevertheless, a significant number of early renal insufficiency patients are also seen to be anaemic.

Most patients in Europe with end stage renal disease are maintained at an Hb level between 6 and 8 mmol/l. According to a survey during the second European Epoetin symposium (Creta, 1998) only 20% is maintained at Hb = 8 mmol/l, but most are maintained at values lower than 8 mmol/l. Even about 40% was maintained at Hb = 6 mmol/l.

A number of studies have found a relationship between left ventricular hypertrophy and haemoglobin in dialysis and pre-dialysis patients. Also a relation between LVH and morbidity and mortality has been found. For this reason it should be a suggestion to treat anaemia towards a higher level.

To treat Hb to a higher level a choice can be made to correct Hb when it has dropped to a very low level after renal disease has reached an advanced stage or alternatively to prevent anaemia in an early stage of renal disease. In an analysis of the normal hematocrit trial, Macdougall and Ritz suggest the latter. This is the main purpose of this trial.

Treatment with Epoetin alfa also makes patients feel better physically when their exercise capacity improves. During treatment with Epoetin alfa, several secondary effects may simultaneously influence the maximal exercise capacity after correction of the anaemia. The improved well-being may result in an increase in physical activity and exercise capacity can be further improved by such conditioning. The improved oxygen transport after correction of anaemia reverses the circulatory adaptation to hypoxia and most studies have shown a decrease in cardiac output at rest, and an increase in peripheral resistance. However, approximately one-third of chronic renal failure patients treated with Epoetin alfa have episodes of hypertension, and may require increased doses of anti-hypertensive medication.

This prospective study will assess whether maintaining Hb levels at normal or sub-normal levels can influence the health status, left ventricular mass and quality of life (QoL) of early renal insufficiency subjects without additional safety concerns. The patients will receive Epoetin Alfa as subcutaneous or intravenous injections in variable dosages for a maximum of 42 months

ELIGIBILITY:
Inclusion Criteria:

* Patients with early renal insufficiency who are not on haemodialysis
* A baseline Hb level of >7.5 mmol/l (120 g/l) but expected to decrease during the coming months. Allowed exceptions: Hb < 7,5 mmol/l (120 g/l) for a maximum of 6 months. In medical history an Hb < 7,0 mmol/l (113 g/l) is only allowed for a maximum period of 3 months and in relation to an accidental drop in Hb (f.e. caused by surgery, gastric bleeding etc.)
* Age: 18 - 73 years, given that patients >70 years are in good general condition and are expected to complete the 30 months study period
* Creatinine clearance < 40 ml/min/1.73 m2 (Cockcroft formula) or creatinin clearance < 50 ml/min/1.73 m2), given that the clearance and Hb show a downward tendency as demonstrated in the patient files and medical history

Exclusion Criteria:

* Presence of clinically significant disease/dysfunction of hepatic, pulmonary, hematological (e.g. sickle cell anaemia, thalassemia, major myelodysplastic syndromes, hemolytic anaemia), neurological, musculo-skeletal, endocrine, gastrointestinal or genitourinary system unrelated to underlying chronic renal failure which in the opinion of the investigator would disqualify the patient from this study
* Cystic kidney disease
* Clinical or laboratory evidence of untreated iron, folate or Vitamin B12 deficiency
* Presence of concomitant malignancy (other than basal cell carcinoma of the skin)
* Uncontrolled hypertension (i.e. diastolic blood pressure of > 100 mm Hg)
* History of seizures
* Administration of medication known to suppress erythropoiesis (e.g. cytotoxic agents, immuno-suppressive) within one month prior to enrolment. Low dose steroid therapy will be permitted
* Pregnancy or lactation
* Known hypersensitivity to Epoetin alfa or one of its components.

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 1999-11; Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Absolute change in left ventricular mass index

SECONDARY OUTCOMES:
Incidence of Left Ventricular hypertrophy QoL assessment (FACIT-Fatigue Scale and KDQOL-SFÒ) The change in pulse pressure during the study period. Morbidity and mortality during the study-period Deterioration of renal function Days in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.